CLINICAL TRIAL: NCT01105104
Title: An Enhanced Medication Monitoring Program
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MedMinder Systems Inc. (Industry)
Collaborators: Narrows Institute for Biomedical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R43HL097395-01A1 (NIH)
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Medication Adherence; Hypertension
MeSH Terms: conditions — Medication Adherence; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MedMinder System (Other)
  Interventions: Device: MedMinder System
- MedMinder System - deactivated (Other)
  Interventions: Device: MedMinder System - deactivated

INTERVENTIONS:
Device: MedMinder System — Participants will receive a fully activated reminder unit as well as at least one call per month from a counselor.
  Arms: MedMinder System
Device: MedMinder System - deactivated — Participants will receive a one-way reminder unit that will remotely transit information on medication adherence
  Arms: MedMinder System - deactivated

SUMMARY:
The goal of the Enhanced Medication Management Program (eMMp) being developed by MedMinder Systems, Inc. is to increase the ability of frail elders to adhere to complex medication regimens for chronic conditions. Adherence will facilitate effective self-care and decrease personal and societal costs associated with disease progression and loss of independence. Multiple studies have shown that more frequent personal follow-up is the most effective way to maximize medication adherence, but such personal care is too costly to translate well to real life in a world of limited healthcare resources.

Currently available "smart pillboxes" are too expensive, too limited in the number and types of medications delivered, and too technically complex for the large majority of senior citizens. The eMMp is designed to deliver prompts and reminders to the user, to be remotely programmable by caregivers, to allow the option of using pre-filled medication trays, to provide electronic adherence reports to family/caregivers and to provide personalized reinforcing phone calls from professional caregivers, all at a modest cost. The in-home ReMinder will use a familiar pillbox layout (4 doses/day for 7 days) and allow easy removal of medication cups by elderly, rheumatic fingers. Installation will require only an electrical outlet (no modems or dedicated phone lines). Once plugged in, the built-in pager will continuously download remotely programmed visual and/or aural prompts and reminders from a central server (RemoteMind). It will continuously upload the date and time when each medi-cation cup is removed and when weekly refill is carried out, enabling remote adherence monitoring, alerts to caregivers, and follow-up intervention(s) from personal and/or professional caregivers as needed.

The hypothesis to be tested in this 2 year SBIR Phase I work plan is that the eMMp will significantly im-prove adherence and clinical outcome (blood pressure control) in a population of frail elderly who are hyper-tensive. SBIR Phase II will determine the minimum level of intervention needed to achieve sustained medication adherence and control of blood pressure in a larger group of hypertensive elders.

ELIGIBILITY:
Inclusion Criteria:

* persons aged 55 years and older who are coming in for routine outpatient visits
* speaks and reads English
* history of high blood pressure
* systolic blood pressure ≥ 130 mm Hg
* using antihypertensive medication
* using 2 or more prescription medications
* plans to stay in area for the 9 months of study

Exclusion criteria:

* receives personal help or reminders to take medication
* has moderate to severe dementia (MMSE score<18)
* has severe hearing or vision deficiency

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-05 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
medication adherence | 6 months
change in systolic blood pressure | 6 months

SECONDARY OUTCOMES:
change in self-efficacy about taking medication | 6 months
self-reported medication taking | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- VA New York Harbor Healthcare System, New York, New York, United States